CLINICAL TRIAL: NCT00572403
Title: Risk Factors Contributing to the Development of Microalbuminuria Over a 5 Year Period
Brief Title: Risk Factors Contributing to the Development of Microalbuminuria
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Responsible Party: Sheldon Tobe, Sunnybrook Health Sciences Centre
Other Study IDs: 298-2007; IISP#P2350
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Microalbuminuria
Keywords: microalbuminuria; risk factors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This research project will look at the relationship between baseline variables, and the new onset of microalbuminuria and the response to treatment with an angiotensin receptor blocker, losartan, in a cohort of 246 early hypertensives and normotensives who are being brought back for a 4-5 year follow up visit as part of a continuing project. We hypothesize that the new onset of microalbuminuria is associated with higher blood pressure levels at baseline and 1 year as well as being associated with elevated left ventricular mass index. The rate of new onset microalbuminuria in non-diabetics is not established and this prospective study will provide data.

DETAILED DESCRIPTION:
The primary objective of this research project is to determine risk factors related to the development of microalbuminuria. The secondary objective is to determine whether uric acid levels at the final visit are correlated with the onset of microalbuminuria. Of participants returning for a 4-5 year follow up visit as part of a continuing project, we will examine the proportion that have developed microalbuminuria. Subjects found to have microalbuminuria will be offered therapy with the ARB losartan and will be followed at three months to determine if there has been a reduction in levels.

ELIGIBILITY:
Inclusion Criteria:

* participation in the Double Exposure study
* elevated microalbuminuria

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants returning for a 4-5 year follow-up visit as part of an ongoing research project will be screened for microalbuminuria and invited to participate if they meet the appropriate criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2007-12; Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
To determine risk factors related to the development of microalbuminuria. | 3 months

SECONDARY OUTCOMES:
To determine whether uric acid levels at the final visit are correlated with the onset of microalbuminuria. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Tobe, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada